CLINICAL TRIAL: NCT07354100
Title: Bifidobacterium Lactulose Optimization in Oncology and Microbiome (BLOOM)
Brief Title: Lactulose to Improve Gut Health in Cancer Patients Receiving Immunotherapy
Acronym: (BLOOM)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB25-1467
Record Dates: First submitted 2026-01-15; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Lactulose

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1 Arm (Experimental): Patients with solid tumor cancers receiving routine immunotherapy will be enrolled to receive lactulose (10 mg daily).
  Interventions: Drug: Lactulose
- Phase 2 Arm (Experimental): o Patients with melanoma receiving routine immunotherapy will be enrolled to receive lactulose (10 mg daily).
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: Lactulose — Lactulose 10 g daily with standard-of-care Immune checkpoint inhibitors (ICIs).

SUMMARY:
The purpose of this study is to see if lactulose can improve the effectiveness of immunotherapy in patients with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria Phase I
* Patients must have a histologically confirmed malignancy that is to receive exclusively ICIs (no chemotherapy or RT in combination) per standard of care during the time in which lactulose will be administered. This includes, but is not limited to, melanoma, cutaneous squamous cell carcinoma, non-small cell lung cancer, mesothelioma, head and neck squamous cell carcinoma, classical Hodgkin lymphoma, primary mediastinal large B-cell lymphoma, urothelial cancer, MSI/MMRd cancer, cancers with high tumor mutational burden (>=10 muts/mB), esophageal cancer, hepatocellular carcinoma, and renal cell carcinoma. Anti-PD-1 or anti-PD-L-1 therapy combinations with anti-LAG-3 or anti-CTLA-4 combinations are permitted.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of lactulose in combination with ICIs in patients <18 years of age, children are excluded from this study.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Patients must be able to ingest liquids.
* Inclusion Criteria Phase II
* Patients must have a histologically confirmed cutaneous or mucosal melanoma. Uveal melanoma is excluded.
* Measurable disease per RECIST 1.1.32
* Documented primary or acquired resistance to anti-PD-1 and anti-CTLA4 therapy per SITC guidelines.21 Primary resistance is defined as disease progression after a minimum of 6 weeks of therapy, provided the patient has received at least two full cycles of treatment, and there has been no prior evidence of clinical benefit (partial response, complete response, or stable disease lasting at least 6 months). Acquired resistance is defined as disease progression after an initial clinical benefit while still on therapy or within 12 weeks of discontinuing therapy, provided the patient received at least two cycles and 6 weeks of therapy.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Planned to receive standard ICI therapy (no RT/ICI or chemotherapy/ICI combinations).
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of lactulose in combination with ICIs in patients <18 years of age, children are excluded from this study.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Patients must be able to ingest liquids.

Exclusion Criteria:

* Exclusion Criteria for Phase I
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ICIs or lactulose.
* Current serious concomitant illnesses include cardiovascular diseases (such as uncontrolled congestive heart failure, hypertension, cardiac ischemia, myocardial infarction, and severe cardiac arrhythmias), bleeding disorders, autoimmune diseases, severe obstructive or restrictive pulmonary diseases, active systemic infections, and inflammatory bowel disorders, including HIV or AIDS-related illnesses or active hepatitis B or C virus.
* The ongoing use of systemic antibiotics or the previous use of antibiotics in the 2 weeks before enrollment.
* Presence of a chronic intestinal disease (for example, celiac, or malabsorption) where the frequency of bowel movements would interfere with study assessments.
* Absence of the large bowel.
* The presence of absolute contraindications to lactulose administration includes galactosemia or other conditions that necessitate a low intake of galactose.
* Expected to require any other form of systemic anti-neoplastic therapy while in the study (i.e., chemotherapy or radiation therapy).
* Symptomatic CNS metastases and/or leptomeningeal involvement. Patients with CNS metastases and/or leptomeningeal involvement may participate if they are clinically stable, as judged by the enrolling investigator.
* Has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo, type I diabetes, or resolved childhood asthma/atopy are exceptions to this rule.
* A history of immune-related adverse events to ICIs that precludes the investigator from comfortably re-challenging with ICIs.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Exclusion Criteria for Phase II
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥ 2 years.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ICIs or lactulose.
* Current serious concomitant illnesses include cardiovascular diseases (such as uncontrolled congestive heart failure, hypertension, cardiac ischemia, myocardial infarction, and severe cardiac arrhythmias), bleeding disorders, autoimmune diseases, severe obstructive or restrictive pulmonary diseases, active systemic infections, and inflammatory bowel disorders, including HIV or AIDS-related illnesses or active hepatitis B or C virus.
* The ongoing use of systemic antibiotics or the previous use of antibiotics in the 2 weeks before enrollment.
* Presence of a chronic intestinal disease (for example, celiac, or malabsorption) where the frequency of bowel movements would interfere with study assessments.
* Absence of the large bowel
* The presence of absolute contraindications to lactulose administration includes galactosemia or other conditions that necessitate a low intake of galactose.
* Expected to require any other form of systemic anti-neoplastic therapy while in the study (i.e., chemotherapy or radiation therapy).
* Symptomatic CNS metastases and/or leptomeningeal involvement. Patients with CNS metastases and/or leptomeningeal involvement may participate if they are clinically stable, as judged by the enrolling investigator.
* Has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo, type I diabetes, or resolved childhood asthma/atopy are exceptions to this rule.
* A history of immune-related adverse events to ICIs that precludes the investigator from comfortably re-challenging with ICIs.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2029-04-13 (Estimated); Study Completion 2029-04-13 (Estimated)

PRIMARY OUTCOMES:
Phase 1- | Baseline to week 3
  Change in Bifidobacterium abundance in stool from baseline to week 3.
Overall Response Rate | Through study completion, an average of 2 years
  Assessment of cancer response based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Phase 1-Safety and tolerability | 3 weeks
  Incidence and severity of adverse events (Common Terminology Criteria for Adverse Events (CTCAE) v5.0) and dose limiting toxicities.
Phase 1- Effects of lactulose | Baseline to week 3
  Change from baseline to week 3 in stool and blood metabolite profiles.
Phase 1- Effects of lactulose | Baseline to week 3
  Change from baseline to week 3 in the abundance of secondary gut microbial taxa and change in alpha diversity indices from baseline to week 3.
Phase 1- Anti-Tumor Evalution | Baseline to week 3
  Evaluating the duration of response, disease control, overall survival, progression free survival and best Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 response.
Phase 2- Safety and tolerability | 12 weeks
  Incidence and severity of adverse events (Common Terminology Criteria for Adverse Events (CTCAE) v5.0) and dose limiting toxicities.
Phase 2- Evaluate changes of stool and serum | Baseline to week 12
  Change from baseline to week 3 in stool and blood metabolite profiles.
Phase 2- Secondary Gut Evaluation | Baseline to week 3
  Change from baseline to week 3 in the abundance of gut microbial tax.
Phase 2- Gut Evaluation | Baseline to week 12
  Change in alpha diversity indices from baseline to week 12.